CLINICAL TRIAL: NCT05555797
Title: Efficacy of Excimer Laser Combined With Either Topical Tazarotene or Topical Betamethasone Valerate Versus Excimer Laser Alone in Treatment of Localized Chronic Plaque Psoriasis; Clinical and Dermoscopic Study
Brief Title: Excimer Laser With Topical Agents in Psoriasis Vulgaris
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliaa Effat Saied Sayed, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXCTBVPS
Record Dates: First submitted 2022-09-17; First posted 2022-09-27 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Lasers, Excimer; Betamethasone Valerate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group of patients with psoriasis vulgaris (Experimental): in each patient lesions will be divided into 3 groups; Group 1: treated with Excimer laser alone(1-2 sessions/ week for 12 sessions according to induration protocol*).
  Group 2: treated with Excimer laser combined with topical tazarotene gel 0.1% Group3: treated with Excimer laser combined with topical betamethasone valerate ointment 0.1%
  Interventions: Device: 308nm Excimer laser; Drug: Tazarotene Topical Gel; Drug: Betamethasone Valerate

INTERVENTIONS:
Device: 308nm Excimer laser — Excimer laser will be (1-2 sessions/ week for 12 sessions according to induration protocol)
Drug: Tazarotene Topical Gel — Tazarotene gel 0.1%(finger tip unit of the gel) will be applied once daily for weeks
Drug: Betamethasone Valerate — .Betamethasone valerate ointment 0.1% will be applied twice daily for 12 weeks.

SUMMARY:
Psoriasis is a chronic, immune-mediated disease that affects approximately 2% of the population. The development and exacerbation of psoriasis involve an interaction between multiple genetic and environmental risk factors.

DETAILED DESCRIPTION:
Psoriasis presents as well-circumscribed, erythematous plaques with an overlying silvery white scales. It has an effect on various aspects of life including mental health, productivity and relationships.

Topical therapies as corticosteroids and vitamin D3 analogs are first-line treatments for mild plaque psoriasis; which involves less than 3% of the body surface area (BSA). Moderate-to-severe plaque psoriasis is usually managed with phototherapy, systemic or biologic therapies .

The American Academy of Dermatology gives a strength recommendation for the use of combination therapies for treatment of psoriasis with superior efficacy to monotherapy .

The 308-nm excimer laser has been widely used for many dermatological diseases. In psoriasis, it shows an efficacy in the treatment of localised plaques especially on the knees and elbows.

It is indicated in moderate to severe psoriasis that affects <10% of the body surface. Areas such as nose, ears and palpebral region can be easily accessed using the laser. It induces lymphocytic apoptosis and decreases the proliferation rate of keratinocytes . There are multiple protocols that evaluate the clinical response to Excimer laser; the induration protocol, the minimal erythema dose and the minimal blistering dose.

The induration protocol compared with the others, allows to modify the dose with treatment. With this protocol, plaques achieved Psoriasis area and severity index (PASI-75) after 10 treatments .

Tazarotene (TAZ) is a topical retinoid with retinoic acid receptor β / γ receptor specificity. It has been shown to be effective for psoriasis treatment. However, its topical application is limited by its irritation.

Studies have shown that combination with other lines may optimize the efficacy as well as minimize the local irritation due to TAZ.

Betamethasone valerate (BV) is a high-potency, synthetic corticosteroid which acts on the intracellular glucocorticoid receptor.

It also binds to membrane-bound receptors, enhancing its action. BV suppresses the production of inflammatory cytokines and reduces keratinocyte hyperproliferation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years.
2. Pattern: Patients with chronic plaque psoriasis not exceeding 10% of the body surface area.

Exclusion Criteria:

1. History of retinoid use either topical or systemic in the previous 16 weeks, phototherapy or topical psoriasis treatment within the last 4 weeks.
2. Allergy to any ingredients of tretinoin or betamethasone drugs.
3. Renal, hepatic disease, cardiovascular , Immunosuppressive therapy, endocrine and blood disease or mental illness.
4. Pregnancy, breast-feeding or women planning to become pregnant within 3 months.
5. Psoriasis exceeding 10% of body surface area or other severe types of psoriasis requiring systemic treatment.
6. Patients with other diseases and requiring treatment that would affect the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-30 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
detection of improvement of psoriasis | 3 months
  detection of improvement of psoriasis in response to excimer laser alone versus its combination with either topical tazarotene gel or betamethasone valerate ointment

SECONDARY OUTCOMES:
dermoscopic role | 3 months
  detection the role of the dermoscope in monitoring the response to treatment of psoriasis by excimer laser alone versus its combination with either topical tazarotene gel or betamethasone valerate ointment.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Abrouk M, Levin E, Brodsky M, Gandy JR, Nakamura M, Zhu TH, Farahnik B, Koo J, Bhutani T. Excimer laser for the treatment of psoriasis: safety, efficacy, and patient acceptability. Psoriasis (Auckl). 2016 Dec 12;6:165-173. doi: 10.2147/PTT.S105047. eCollection 2016. PMID 29387603
- [Result] Ardeleanu V, Sabina Radaschin D, Tatu AL. Excimer laser for psoriasis treatment: A case report and short review. Exp Ther Med. 2020 Jul;20(1):52-55. doi: 10.3892/etm.2020.8529. Epub 2020 Feb 14. PMID 32508993
- [Result] He C, Jin H, Liu X, Hu F, Zhang L, Zhang S, He Y, Yang X, Chen H, Wang X, Ji C, Lv C, Miao G, Li X, Diao Q, Li L, Li X, Li Y, Wang R, Zhang L, Zhou X, Xia X, Yan M, Song J, Zhang R, Geng L, Zheng M, Lu Q, Lu T, Shi Y, Jing H, Zhang X, Shi J, Xia J, Gao Y, Wang Y. Tazarotene/Betamethasone Dipropionate Cream in Patients with Plaque Psoriasis: Results of a Prospective, Multicenter, Observational Study. Dermatology. 2021;237(4):603-610. doi: 10.1159/000511891. Epub 2020 Dec 22. PMID 33352561
- [Result] Elmets CA, Korman NJ, Prater EF, Wong EB, Rupani RN, Kivelevitch D, Armstrong AW, Connor C, Cordoro KM, Davis DMR, Elewski BE, Gelfand JM, Gordon KB, Gottlieb AB, Kaplan DH, Kavanaugh A, Kiselica M, Kroshinsky D, Lebwohl M, Leonardi CL, Lichten J, Lim HW, Mehta NN, Paller AS, Parra SL, Pathy AL, Siegel M, Stoff B, Strober B, Wu JJ, Hariharan V, Menter A. Joint AAD-NPF Guidelines of care for the management and treatment of psoriasis with topical therapy and alternative medicine modalities for psoriasis severity measures. J Am Acad Dermatol. 2021 Feb;84(2):432-470. doi: 10.1016/j.jaad.2020.07.087. Epub 2020 Jul 30. PMID 32738429
- [Result] Nestor MS, Fischer D, Arnold D. Randomized, Investigator-Blinded Study to Compare the Efficacy and Tolerance of a 650-microsecond, 1064-nm YAG Laser to a 308-nm Excimer Laser for the Treatment of Mild to Moderate Psoriasis Vulgaris. J Drugs Dermatol. 2020 Feb 1;19(2):176-183. doi: 10.36849/JDD.2020.4769. PMID 32129962
- [Result] Langley RG, Ellis CN. Evaluating psoriasis with Psoriasis Area and Severity Index, Psoriasis Global Assessment, and Lattice System Physician's Global Assessment. J Am Acad Dermatol. 2004 Oct;51(4):563-9. doi: 10.1016/j.jaad.2004.04.012. PMID 15389191
- [Result] Ramez SA, Soliman MM, Fadel M, Nour El-Deen F, Nasr M, Youness ER, Aboel-Fadl DM. Novel methotrexate soft nanocarrier/fractional erbium YAG laser combination for clinical treatment of plaque psoriasis. Artif Cells Nanomed Biotechnol. 2018;46(sup1):996-1002. doi: 10.1080/21691401.2018.1440236. Epub 2018 Feb 15. PMID 29448838
- [Result] Taneja A, Trehan M, Taylor CR. 308-nm excimer laser for the treatment of psoriasis: induration-based dosimetry. Arch Dermatol. 2003 Jun;139(6):759-64. doi: 10.1001/archderm.139.6.759. PMID 12810507
- [Result] Naldi L, Yawalkar N, Kaszuba A, Ortonne JP, Morelli P, Rovati S, Mautone G. Efficacy and safety of the Betamethasone valerate 0.1% plaster in mild-to-moderate chronic plaque psoriasis: a randomized, parallel-group, active-controlled, phase III study. Am J Clin Dermatol. 2011 Jun 1;12(3):191-201. doi: 10.2165/11539780-000000000-00000. PMID 21284407